CLINICAL TRIAL: NCT03011775
Title: Effect of Pioglitazone on Insulin Resistance, Progression of Atherosclerosis and Clinical Course of Coronary Heart Disease
Brief Title: Effect of Pioglitazone on Insulin Resistance, Atherosclerosis Progression and Clinical Course of Coronary Heart Disease
Acronym: EFFORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ukrainian Medical Stomatological Academy (Other)
Responsible Party: Principal Investigator, Igor Kaydashev, Head of Internal Medicine Department #3, Ukrainian Medical Stomatological Academy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT-18-06-2012
Record Dates: First submitted 2016-12-29; First posted 2017-01-05 (Estimated); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-01

CONDITIONS: Adverse Effect; Atherosclerosis, Coronary; Insulin Resistance Syndrome
Keywords: Pioglitazone, Insulin Resistance; Atherosclerosis, Coronary Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Metabolic Syndrome; Insulin Resistance; Atherosclerosis; Coronary Disease | interventions — Pioglitazone; Tablets; Hypoglycemic Agents; Isosorbide Dinitrate; Vasodilator Agents; Aspirin; Anti-Inflammatory Agents, Non-Steroidal; Platelet Aggregation Inhibitors; Bisoprolol; Rosuvastatin Calcium; Hypolipidemic Agents; Ramipril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone + Standard Care (Experimental): 20 patients who received standard medical therapy complex: isosorbide dinitrate 10-20 mg 2 times a day, acetylsalicylic acid 75 mg 1 time a day, bisoprolol 2.5 mg 1 time a day, rosuvastatin 20 mg 1 time a day, ramipril 5 mg 1 time a day. Patients also received recommendations on diet and lifestyle changes. Included pioglitazone 15 mg 1 time per day in the morning for 6 months.
  Interventions: Drug: Pioglitazone 15 mg Tablet; Drug: Isosorbide Dinitrate 10Mg Tablet; Drug: Acetylsalicylic Acid 75Mg Tablet; Drug: Bisoprolol Fumarate 2.5 MG Oral Tablet; Drug: Rosuvastatin Calcium 20 MG Oral Tablet; Drug: Ramipril 5 MG
- Standard Care (Other): 23 patients who received standard medical therapy complex: isosorbide dinitrate 10-20 mg 2 times a day, acetylsalicylic acid 75 mg 1 time a day, bisoprolol 2.5 mg 1 time a day, rosuvastatin 20 mg 1 time a day, ramipril 5 mg 1 time a day. Patients also received recommendations on diet and lifestyle changes.
  Interventions: Drug: Isosorbide Dinitrate 10Mg Tablet; Drug: Acetylsalicylic Acid 75Mg Tablet; Drug: Bisoprolol Fumarate 2.5 MG Oral Tablet; Drug: Rosuvastatin Calcium 20 MG Oral Tablet; Drug: Ramipril 5 MG

INTERVENTIONS:
Drug: Pioglitazone 15 mg Tablet — Pioglar (Ranbaxy India):1 tablet per day in the morning for 6 months
  Other Names: Oral hypoglycemic agent
  Arms: Pioglitazone + Standard Care
Drug: Isosorbide Dinitrate 10Mg Tablet — 1-2 tablets 2 times a day
  Other Names: Antianginal, vasodilator agent
Drug: Acetylsalicylic Acid 75Mg Tablet — 1 tablet per a day
  Other Names: NSAID and antiplatelet agent
Drug: Bisoprolol Fumarate 2.5 MG Oral Tablet — 1 tablet per a day
  Other Names: Lowering high blood pressure agent
Drug: Rosuvastatin Calcium 20 MG Oral Tablet — 1 tablet per a day
  Other Names: Lipid- lowering agent
Drug: Ramipril 5 MG — 1 tablet per a day
  Other Names: ACE inhibitor

SUMMARY:
Pioglitazone, a medication of thiazolidinedione group, is capable of triggering the peroxisome proliferator-activated receptors (PPAR-γ). Activation of receptor PPAR-γ regulates carbohydrate and lipid metabolism, immune and inflammatory responses in heart tissues.

Our aim will to study the effect of pioglitazone on insulin resistance, the clinical course of atherosclerosis and coronary heart disease (CHD).

The study will include 43 patients with coronary artery disease. Patients will be divided into the study group - 20 patients, in whom pioglitazone will be included in the combined therapy at a dose of 15 mg 1 time per day in the morning, and the control group - 23 patients receiving standard complex drug therapy over 6 months. Patients will be underwent clinical examination, ultrasound of neck vessels, study of carbohydrate and lipid metabolism.

The end primary points of the study will be the onset of death due to myocardial infarction, coronary revascularization procedures (coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI)), or hospitalization for acute coronary syndrome (ACS) or unstable angina (UA).

Predefined secondary end points included carotic atherosclerotic leisure (carotic intima-media thickness, diameter of stenosis, presents of atherosclerotic plaque), systemic inflammation level (the level of C reactive protein), lipid metabolism (levels of serum total cholesterol, triglycerides, high and low density lipoproteins), level of insulin resistance ( oral glucose tolerance test, blood glucose).

DETAILED DESCRIPTION:
The study will include 43 people aged between 45 and 68 who suffered from ischemic heart disease. Before starting the study, all participants will give written informed consent, will be obtained of the Commission on Bioethics at Ukrainian Medical Stomatological Academy. Inclusion criteria will be as follows: stable exertional angina, type 2 diabetes mellitus (DM) without receiving injectable antidiabetic drugs. Exclusion criteria will be: the presence of myocardial infarction history, intervention, malignant arterial hypertension (AH), chronic heart failure (HF) of III-IV functional class (FC), systemic connective tissue diseases, cancer and oncohematological diseases, severe infectious diseases, chronic inflammatory diseases, history of acute cerebrovascular accidents, disorders of cardiac rhythm by atrial fibrillation type. The end study will be the primary points: the onset of death due to myocardial infarction, coronary revascularization procedures (coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI)), or hospitalization for acute coronary syndrome (ACS) or unstable angina (UA).

The diagnosis of CHD in patients will confirmed by the presence of FC I-III angina according to the classification of the Canadian Cardiovascular Society and the phenomena of circulatory insufficiency according to the classification of New York Heart Association (NYHA). Bicycle ergometry will perform on "Veloergotest 05" (Ukraine) via step increasing loading capacity with a consequent increase under control of electrocardiogram (ECG) and BP. The force of step I will be 150 kgm / min (25 W); II - 300 kgm / min (50 W); III - 450 kgm / min (75 W); IV - 600 kgm / min (100 W); V - 750 kgm / min (125 W); VI - 900 kgm / min (150 W), the duration of each step was 3 minutes. Tolerance of CHD patients to exercise will calculate from the value of the threshold load capacity and volume of work performed. The threshold load capacity of 150 kgm / min (25 W) was considered very low and consistent with angina FC IV; 300 kgm / min (50 W) - low, FC III; 450-600 kgm / min (75-100 W) - average, FC II; 750 kgm / min (125 W) and above - high exercise capacity, FC I. The criteria will cease bicycle ergometry termination conventional clinical or ECG signs of myocardial ischemia.

Prior to inclusion in the clinical trial, all patients will receive conventional treatment and will screening examination to verify the diagnosis of coronary heart disease and type 2 diabetes.

After screening, we will selected 43 patients who received standard medical therapy complex: isosorbide dinitrate 10-20 mg 2 times a day, acetylsalicylic acid 75 mg 1 time a day, bisoprolol 2.5 mg 1 time a day, rosuvastatin 20 mg 1 time a day, ramipril 5 mg 1 time a day. Patients also will receive recommendations on diet and lifestyle changes. Patients will receive the conventional treatment for at least one month to achieve stable parameters.

On the first day of the study, blood samples will take from all patients, clinical examination was conducted. After clinical and laboratory studies, patients will randomized by gender, age and severity of clinical manifestations of coronary heart disease. As a result of randomization, patients will divide into the study group (n = 20) and control group (n = 23). The complex therapy of the study group will include pioglitazone 15 mg 1 time per day in the morning ("Pioglar", Ranbaxy, India) for 6 months. Patients of the control group will continue to receive only a standard set of drug therapy. Re-examination will carry out in 6 months.

The examination will include the collection of medical history and objective data (gender, age, overweight and obesity, hypertension, type 2 diabetes). Patients will evaluate by anthropometric indicators (height, weight, body mass index (BMI)), blood pressure - systolic and diastolic (SBP and DBP), heart rate (HR) will measure, ECG will register.

In order to determine the status of vascular bed, patients will underwent ultrasonography (US) of neck vessels on "ULTIMA PA", sensor L5 - 12/40, in accordance with standard protocols in B-mode on the three levels of vascular bed and bilaterally at the end of diastole: in the proximal, medial and distal points at a distance of 1 cm from the bifurcation of the posterior wall of the right and left common carotid artery (RCCA and LCCA, respectively) as more distant from the transducer unit. Contour of the carotid arteries will register, their inner lumen, indicators for ASP presence (size, localization) will record, as well as IMT of the carotid arteries. IMT will measure as the distance between the first and the second echogenic lines of located site according to the procedure Pignoli P. et al. The diameter of RCCA, LCCA, and the internal carotid artery (ICA) will assess at the end of systole and diastole as the distance between the IMT. Normal IMT will consider less than 0.9 mm; CCA IMT > 1.4 mm was evaluated as ASP, and in the range of 1.0-1.3 mm as the thickening of IMT (ESH, ESC, 2007). The standard criteria for the diagnosis of hemodynamically significant stenosis are the narrowing of the arterial lumen by more than 50%.

The volume of laboratory tests will includ general clinical and biochemical blood analysis. For the control of carbohydrate metabolism glycemic profiles will study determining fasting glucose and after 1 hour after taking 75 g of glucose (oral glucose tolerance test, OGTT) via glucose oxidase method; hyperglycemic factor will calculate. In all patients lipid profile will studied: total cholesterol (TC), triglycerides (TG) and cholesterol of high-density lipoproteins (HDL) ("Diakon-DS", Russia), content of cholesterol in low-density lipoproteins (LDL) and very low density lipoproteins (VLDL) will calculate, as well as atherogenic factor (AF). Study of the inflammatory response will conduct by determining the concentration of basic biomarkers - high-sensitivity C-reactive protein (hs-CRP, "DRG", USA), human tissue inhibitor of metalloproteinase-1 (TIMP-1, "eBioscience", Austria) according to the manufacturer's protocols of test systems via immunoenzyme method. The presence of microalbuminuria will determine using test strips "Mikroalbufan" ("Lachema", Czech Republic), the ratio albumin / creatinine in urine will calculated.

Statistical processing will perform using software "Statistica 6.0" (StatSoft, USA) with calculation of average (M) and standard error of the average (m). Methods of descriptive statistics will use, comparison of performance in groups will perform by parametric (Student's t-test) and non-parametric (Pearson χ2 test, Fisher's exact test, Mann-Whitney test) statistics. For all types of analysis the differences at p <0.05 will consider statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* stable exertional angina,
* type 2 diabetes mellitus (DM) without receiving injectable antidiabetic drugs

Exclusion Criteria:

* the presence of myocardial infarction history, intervention;
* malignant arterial hypertension (AH);
* chronic heart failure (HF) of III-IV functional class (FC);
* systemic connective tissue diseases;
* cancer and oncohematological diseases, severe infectious diseases, chronic inflammatory diseases;
* history of acute cerebrovascular accidents;
* disorders of cardiac rhythm by atrial fibrillation type.

Ages: 45 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ukrainian Medical Stomatological Academy, Poltava, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Struijker Boudier HA, Zanchetti A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Kjeldsen SE, Erdine S, Narkiewicz K, Kiowski W, Agabiti-Rosei E, Ambrosioni E, Cifkova R, Dominiczak A, Fagard R, Heagerty AM, Laurent S, Lindholm LH, Mancia G, Manolis A, Nilsson PM, Redon J, Schmieder RE, Struijker-Boudier HA, Viigimaa M, Filippatos G, Adamopoulos S, Agabiti-Rosei E, Ambrosioni E, Bertomeu V, Clement D, Erdine S, Farsang C, Gaita D, Kiowski W, Lip G, Mallion JM, Manolis AJ, Nilsson PM, O'Brien E, Ponikowski P, Redon J, Ruschitzka F, Tamargo J, van Zwieten P, Viigimaa M, Waeber B, Williams B, Zamorano JL, The task force for the management of arterial hypertension of the European Society of Hypertension, The task force for the management of arterial hypertension of the European Society of Cardiology. 2007 Guidelines for the management of arterial hypertension: The Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). Eur Heart J. 2007 Jun;28(12):1462-536. doi: 10.1093/eurheartj/ehm236. Epub 2007 Jun 11. No abstract available. PMID 17562668

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone + Standard Care: 20 patients who received standard medical therapy complex: isosorbide dinitrate 10-20 mg 2 times a day, acetylsalicylic acid 75 mg 1 time a day, bisoprolol 2.5 mg 1 time a day, rosuvastatin 20 mg 1 time a day, ramipril 5 mg 1 time a day. Patients also received recommendations on diet and lifestyle changes. Included pioglitazone 15 mg 1 time per day in the morning for 6 months.
  Pioglitazone 15 mg Tablet: 1 tablet per day in the morning for 6 months
  Isosorbide Dinitrate 10Mg Tablet: 1-2 tablets 2 times a day
  Acetylsalicylic Acid 75Mg Tablet: 1 tablet per a day
  Bisoprolol Fumarate 2.5 MG Oral Tablet: 1 tablet per a day
  Rosuvastatin Calcium 20 MG Oral Tablet: 1 tablet per a day
  ramipril 5 MG: 1 tablet per a day
Period: Overall Study
Arm/Group | Pioglitazone + Standard Care | Standard Care
Started | 20 | 23
Completed | 20 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone + Standard Care | Standard Care | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 22 | 41
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (1.15) | 53 (1.36) | 53.7 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 12 | 16 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 23 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Ukraine | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Сardiovascular Death
Description: Number of Participants with cardiovascular death
Time Frame: Baseline and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
Participants
  Baseline | 0 | 0
  1 year | 0 | 0

2. Primary Outcome: Coronary Artery Bypass [Coronary Revascularization]
Description: Number of Participants with revascularization coronary procedures (coronary artery bypass grafting)
Time Frame: Baseline and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
Participants
  Baseline | 0 | 0
  1 year | 0 | 0

3. Primary Outcome: Cardiovascular Hospitalization
Description: Number of Participants with acute coronary syndrome (ACS) or unstable angina (UA)
Time Frame: Baseline and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
Participants
  Baseline | 0 | 0
  1 year | 0 | 0

4. Primary Outcome: Percutaneous Coronary Intervention [Coronary Revascularization]
Description: Number of Participants with incidence of percutaneous coronary intervention.
Time Frame: Baseline and 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Pioglitazone + Standard Care: 20 patients who received standard medical therapy complex: isosorbide dinitrate 10-20 mg 2 times a day, acetylsalicylic acid 75 mg 1 time a day, bisoprolol 2.5 mg 1 time a day, rosuvastatin 20 mg 1 time a day, ramipril 5 mg 1 time a day. Patients also received recommendations on diet and lifestyle changes. Included pioglitazone 15 mg 1 time per day in the morning for 6 months.
  Pioglitazone 15 mg Tablet: 1 tablet per day in the morning for 6 months
  Isosorbide Dinitrate 10Mg Tablet: 1-2 tablets 2 times a day
  Acetylsalicylic Acid 75Mg Tablet: 1 tablet per a day
  Bisoprolol Fumarate 2.5 MG Oral Tablet: 1 tablet per a day
  Rosuvastatin Calcium 20 MG Oral Tablet: 1 tablet per a day
  ramipril 5 MG: 1 tablet per a day
  During the observation of mortality from all-cause mortality, serious adverse events, other (Not Including Serious) adverse events among patients of study groups not recorded.
- Standard Care: 23 patients who received standard medical therapy complex: isosorbide dinitrate 10-20 mg 2 times a day, acetylsalicylic acid 75 mg 1 time a day, bisoprolol 2.5 mg 1 time a day, rosuvastatin 20 mg 1 time a day, ramipril 5 mg 1 time a day. Patients also received recommendations on diet and lifestyle changes.
  Isosorbide Dinitrate 10Mg Tablet: 1-2 tablets 2 times a day
  Acetylsalicylic Acid 75Mg Tablet: 1 tablet per a day
  Bisoprolol Fumarate 2.5 MG Oral Tablet: 1 tablet per a day
  Rosuvastatin Calcium 20 MG Oral Tablet: 1 tablet per a day
  ramipril 5 MG: 1 tablet per a day During the observation of mortality from all-cause mortality, serious adverse events, other (Not Including Serious) adverse events among patients of control groups not recorded.
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
Participants
  Baseline | 0 | 0
  1 year | 0 | 0

5. Primary Outcome: Safety and Tolerability 1
Description: Liver injury: mean values of ALT
Time Frame: Baseline, 6 month and 1 year
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
units per liter (U/L)
  Baseline | 23.4 (2.4) | 26.9 (2.57)
  Mean values of ALT in 6 months | 27.4 (2.1) | 26.1 (1.68)
  Mean values of ALT in 1 year | 19.9 (1.9) | 23.9 (1.19)

6. Primary Outcome: Safety and Tolerability 2
Description: Liver injury: mean levels of total bilirubin
Time Frame: Baseline, 6 month and 1 year
Measure: Mean (Standard Deviation); unit: μmol/l
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
μmol/l
  Baseline | 12.3 (1.3) | 10.8 (1.01)
  Mean values of total bilirubin in 6 month | 12.4 (1.02) | 12.7 (1.05)
  Mean values of total bilirubin in 1 year | 15.7 (1.6) | 15.0 (5.9)

7. Primary Outcome: Safety and Tolerability 3
Description: Kidney injury: mean values of the microalbuminuria
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: mg/mol
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
mg/mol
  Baseline | 31.44 (4.28) | 41.1 (4.85)
  1 year | 31.10 (5.00) | 37.70 (4.48)

8. Primary Outcome: Safety and Tolerability 4
Description: Kidneys injury: mean values of creatinine
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: μmol/l
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
μmol/l
  Mean values of creatinine in men baseline | 105.6 (38.5) | 102.3 (43.1)
  Mean values of creatinine in men in 1 year | 85.0 (21.1) | 82.0 (14.0)
  Mean values of creatinine in women baseline | 66.8 (8.8) | 88.2 (11.1)
  Mean values of creatinine in women in 1 year | 72.5 (8.1) | 77.5 (18.0)

9. Secondary Outcome: Thickness of the Intima-media Complex
Description: Mean thickness of carotid intima-media complex
Time Frame: Baseline, 6 month and 1 year
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
cm
  Mean thickness of the right carotid intima-media baseline | 1.08 (0.17) | 0.98 (0.15)
  Mean thickness of the right carotid intima-media in 6 month | 1.05 (0.13) | 0.97 (0.11)
  Mean thickness of the right carotid intima-media in 1 year | 1.01 (0.02) | 1.01 (0.01)
  Mean thickness of the left carotid intima-media baseline | 1.1 (0.18) | 1.0 (0.15)
  Mean thickness of the left carotid intima-media in 6 month | 1.06 (0.13) | 1.00 (0.10)
  Mean thickness of the left carotid intima-media in 1 year | 1.02 (0.02) | 0.97 (0.02)
Statistical Analysis 1: Comparison: Pioglitazone + Standard Care vs Standard Care; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); The threshold for statistical significance was P value of .05

10. Secondary Outcome: Diameter of Stenosis [Carotic Atherosclerotic Lesions]
Description: Mean diameters of the stenosis of the right and left common carotid arteries
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
mm
  Mean diameter of the stenosis of the right common carotid artery baseline | 9.8 (3.1) | 8.7 (2.7)
  Mean diameter of the stenosis of the right common carotid artery in 1 year | 5.0 (1.8) | 4.8 (1.5)
  Mean diameter of the stenosis of the left common carotid artery baseline | 11.6 (3.6) | 10.1 (3.0)
  Mean diameter of the stenosis of the left common carotid artery in 1 year | 4.1 (1.7) | 5.6 (1.8)
Statistical Analysis 1: Comparison: Pioglitazone + Standard Care vs Standard Care; Test type: Superiority; p > 0.05, Chi-squared

11. Secondary Outcome: Carotic Atherosclerotic Lesions
Description: Number of Participants with presence of atherosclerotic plaque of the intima media of common carotid artery greater than 1.4 mm
Time Frame: Baseline and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
Participants
  Baseline | 0 | 0
  1 year | 0 | 0

12. Secondary Outcome: Systemic Inflammation Level
Description: Number of Participants with C-reactive protein level above 3 mg/L
Time Frame: Baseline and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
Participants
  Baseline | 10 | 7
  In 1 year | 12 | 13
Statistical Analysis 1: Comparison: Pioglitazone + Standard Care vs Standard Care; Test type: Superiority; p > 0.05, Chi-squared

13. Secondary Outcome: Lipid Metabolism 1
Description: Mean levels of total serum cholesterol
Time Frame: Baseline, 6 month and 1 year
Measure: Mean (Standard Deviation); unit: mmol / l
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
mmol / l
  Mean values of the total cholesterol level baseline | 5.27 (0.2) | 5.28 (1.0)
  Mean values of the total cholesterol level in 6 month | 4.5 (0.2) | 4.3 (0.2)
  Mean values of the total cholesterol level in 1 year | 4.5 (0.2) | 4.3 (0.2)
Statistical Analysis 1: Comparison: Pioglitazone + Standard Care vs Standard Care; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Lipid Metabolism 2
Description: Mean values of the triglyceride levels
Time Frame: Baseline, 6 month and 1 year
Measure: Mean (Standard Deviation); unit: 1 mmol/L
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
1 mmol/L
  Mean values of triglyceride baseline | 0.69 (0.1) | 0.61 (0.21)
  Mean values of triglyceride in 6 month | 0.72 (0.40) | 0.73 (0.25)
  Mean values of triglyceride in 1 year | 0.9 (0.1) | 0.7 (0.1)

15. Secondary Outcome: Lipid Metabolism 3
Description: Lipoproteine fractions:mean values of high-density lipoproteins and low density lipoproteins
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
mmol/L
  Mean values of high-density lipoproteins in men baseline | 0.8 (0.2) | 0.9 (0.4)
  Mean values of high-density lipoproteins in men in 1 year | 1.1 (0.3) | 1.0 (0.3)
  Mean values of high-density lipoproteins in women baseline | 0.9 (0.3) | 1.1 (0.2)
  Mean values of high-density lipoproteins in women in 1 year | 1.2 (0.2) | 1.0 (0.2)
  Mean values of low density lipoproteins in men baseline | 3.9 (0.7) | 4.4 (0.8)
  Mean values of low density lipoproteins in men in 1 year | 2.9 (0.5) | 3.0 (0.6)
  Mean values of low density lipoproteins in women baseline | 4.5 (0.8) | 3.5 (0.8)
  Mean values of low density lipoproteins in women in 1 year | 3.3 (0.8) | 2.7 (0.3)
Statistical Analysis 1: Comparison: Pioglitazone + Standard Care vs Standard Care; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

16. Other Pre Specified Outcome: Level of Insulin Resistance 1
Description: Oral glucose tolerance test: number of Participants with impaired glucose tolerance
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
Participants
  Number of Participants with glucose level in the range of 7.8 to 11 mmol/L baseline | 7 | 14
  Number of Participants with glucose level in the range of 7.8 to 11 mmol/L in 6 month | 13 | 16
  Number of Participants with glucose level above 11 mmol/L baseline | 10 | 4
  Number of Participants with glucose level above 11 mmol/L in 6 month | 5 | 3
Statistical Analysis 1: Comparison: Pioglitazone + Standard Care vs Standard Care; Test type: Superiority; p < 0.05, Chi-squared

17. Other Pre Specified Outcome: Level of Insulin Resistance 2
Description: Mean levels of blood glucose
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone + Standard Care | Standard Care
Number analyzed (Participants) | 20 | 23
mmol/L
  Baseline | 6.0 (0.1) | 5.9 (0.54)
  In 6 month | 5.97 (0.20) | 5.60 (0.79)
Statistical Analysis 1: Comparison: Pioglitazone + Standard Care vs Standard Care; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pioglitazone + Standard Care | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 0/20 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes